CLINICAL TRIAL: NCT07346950
Title: The Effect of Autoreactive Autoantibodies on Peripheral and Central Disease Mechanisms in Fibromyalgia.
Acronym: FINE
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-03464-01
Record Dates: First submitted 2025-12-03; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: cytokines; neuroinflammation; blood-brain barrier; BBB; fMRI; autoantibodies; skin; MRS; cerebrospinal fluid
MeSH Terms: conditions — Fibromyalgia; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin (4mm punch biopsy) Serum Plasma Peripheral blood mononuclear cells Cerebrospinal fluid cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FM: Participants with fibromyalgia according to the ACR 1990+2016 criteria.
- HC: Control participants that have no pain condition. No cerebrospinal fluid was collected from this cohort.
- CSF controls: A cohort consisting of 1) healthy controls (n = 11) recruited in another study and 2) patients with non-inflammatory neurological symptoms (NINS, n = 32) that underwent clinical workup at the neurological clinic at Uppsala University Hospital.

SUMMARY:
This observational study aims to compare disease burden and pain characteristics between fibromyalgia patients with high levels of autoreactive autoantibodies, fibromyalgia patients with low levels of autoreactive autoantibodies, and healthy controls. The primary hypothesis is that patients experience more symptoms (as measured with questionnaires) depending on their antibody titer, and that high levels of autoantibodies correlate with other biological markers, such as inflammatory profile in serum, and density of intraepidermal nerve fibers in skin.

The secondary aim of this study is to characterize central markers of disease, which will be done using a number of methods: the investigators will quantify immune profile in the cerebrospinal fluid, measure thalamic neurotransmitter levels with magnetic resonance spectroscopy (MRS), blood-brain barrier permeability with both biochemical markers and T1-weighed gadolinium-enhanced magnetic resonance imaging (MRI), and resting state activity of the brain (MRI). The investigators hypothesize that there are signs of upregulation of the immune system of the central compartment, and that this will be correlated with altered neurotransmitter levels and an altered resting state activity.

ELIGIBILITY:
Inclusion criteria:

* Female sex
* Age 20-70
* Fibromyalgia according to the ACR 1990+2016 criteria for the FM cohort.

Exclusion Criteria:

* Reported BMI > 35 during screening over a phone call.
* Other dominant chronic pain states.
* Autoimmune diseases (exception: primary hypothyroidism).
* Serious somatic or psychiatric disease.
* Current pregnancy.
* Non-fluency in Swedish.
* For HC: history of chronic pain or current pain exceeding 20 on a 0-100 scale or having received an FM diagnosis.
* For NINS: having received an FM diagnosis.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total, 80 subjects with fibromyalgia (FM) and 42 healthy controls (HC) will be included. Subjects predominantly live in Uppsala County, Sweden, which has a population of approximately 400,000 inhabitants. If we consider the prevalence of FM to be 2%, that translates to ~8,000 patients. Since the study is on female subjects, and about 70% of FM patients are female, that leaves about 5,600 patients in the pool. The sample size has been determined based on previous research where a group size of 40 subjects was deemed sizeable enough to identify meaningful differences in expression of proteins. As we are interested in two groups of FM patients, i.e., those with high and low levels of autoreactive autoantibodies, and we expect about 50% of participants with FM to have high titers, we will require about 80 participants in the FM group.
  For the NINS cohort, the biobank of the neurological clinic at Uppsala University Hospital will be utilized to find appropriate CSF controls.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Anti-SGC antibodies | At study inclusion.
  Autoantibodies that bind to satellite glia cells in the dorsal root ganglia. The investigators hypothesize that autoantibody titers are associated with symptom severity (Goebel et al., 2021; Krock et al., 2023; Fanton et al., 2023), changes in inflammatory profile (af Ekenstam et al., 2025) and alterations in skin histological findings.

SECONDARY OUTCOMES:
Neurotransmitter levels in the right thalamus | At study inclusion.
  Using magnetic resonance spectroscopy, the first 55 FM subjects and the first 25 HC subjects had their levels of neurotransmitters in the right thalamus quantified. The investigators hypothesize that FM patients will have upregulated glutamate levels in their thalamus, and that glutamate levels will be associated with restless legs symptom severity.
Inflammatory profile in serum | At study inclusion.
  Using multiplexed proximity-extension assays (OLINK, Uppsala, Sweden), the investigators aim to quantify the levels of cytokines and chemokines in the serum of patients with fibromyalgia and in healthy, pain-free controls. FM patients are hypothesized to have an upregulation of cytokines related to B-cell activity, such as CD40 (af Ekenstam et al., 2025).
Inflammatory profile in cerebrospinal fluid | At study inclusion.
  Using multiplexed proximity-extension assays, the investigators aim to quantify the levels of cytokines and chemokines in the cerebrospinal fluid of patients with fibromyalgia and in control samples from patients that underwent a neurological work-up at the neurological clinic of Uppsala University Hospital. The investigators hypothesize that fibromyalgia patients have upregulated cytokine levels in CSF (Rosenström et al., 2024a), especially regarding e.g. fractalkine, IL8, CCL19, CCL25 - which have previously been found to be upregulated (Bäckryd et al., 2017) and separately been associated with glia cell activity (Maciejewski-Lenoir et al., 1999), BBB permeability (García-Fernández et al., 2023) and fatigue (Rosenström et al., 2025).
CSF-serum albumin quotients | At study inclusion.
  The CSF/serum albumin quotient is the gold standard for quantification of blood-brain barrier integrity. The investigators hypothesize that (female) FM patients will have a more permeable BBB, i.e., higher CSF/serum albumin quotient than (female) patients with lumbar disc herniation, degenerative disc disease, osteoarthritis or control patients, suggesting an increased peripheral-central communication, which in turn has been reported to be important for the central immunoenvironment (Rosenström et al., 2025).
Quantitative sensory testing (QST) | At study inclusion.
  QST was used to measure pressure pain thresholds (PPTs), temporal summation and conditioned pain modulation in all FM and HC subjects. FM are expected to have lower PPTs, a stronger temporal summation and impaired descending inhibition compared to HC (Kosek & Hansson, 1997).
Intraepidermal nerve fiber density (IENFD) in skin | At study inclusion.
  All FM and HC participants gave two 4mm punch biopsies of the skin from their right thigh (lateral). These samples will be used to quantify IENFD to be used as a correlation measure with autoantibody titers and inflammatory profiles in serum. The investigators expect reduced IENFD in patients with fibromyalgia (Üçeyler et al., 2013; Evdokimov et al., 2019), and hypothesize that IENFD will be correlated with autoantibody titers.
Polysomnography | At study inclusion.
  All FM and HC subjects underwent a one-night ambulatory polysomnography to characterize their sleep quality objectively. The investigators hypothesize that fibromyalgia patients have disturbed overall sleep quality (Muza et al., 2023).
Resting state functional magnetic resonance imaging (rsfMRI) | At study inclusion.
  Using rsfMRI, the resting state activity of the brain will be measured in the first 55 FM subjects and in the first 25 HC subjects. We expect a higher functional connectivity in areas related to the default network and lower functional connectivity in areas related to endogenous pain modulation (Cavicchioli et al., 2025).
Blood-brain barrier dynamics | At study inclusion.
  Using a gadolinium-enhanced, T1-weighted MRI method, the investigators will assess the dynamic permeability of the BBB in the brain of the first 55 FM subjects and the first 25 HC subjects. The investigators hypothesize that FM patients will have a more leaky BBB than controls, as indicated by a faster uptake of gadolinium in the CSF and brain parenchyme. This will be quantified by MRI physicists using standard quantification metrics that mirror physiological function.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kosek, MD, PhD, Principal Investigator — Uppsala University, Karolinska Institutet
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden